CLINICAL TRIAL: NCT00151047
Title: Evaluation of Primary Chemotherapy With Docetaxel Plus Capecitabine in Selected Patients With Newly Diagnosed Localized or Locally Advanced Prostate Cancer
Brief Title: Docetaxel Plus Capecitabine in Newly Diagnosed Localized or Locally Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2-42
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel and Capecitabine (Experimental)
  Interventions: Drug: Capecitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Capecitabine
Drug: Docetaxel

SUMMARY:
Purpose: The purpose of this clinical trial is to look at the chemotherapy combination of docetaxel and capecitabine in the treatment of newly diagnosed or locally advanced prostate cancer, and to determine if this treatment is an acceptable, effective and a safe treatment option. In addition, this clinical trial will evaluate how this treatment affects chemicals (enzymes), and other cancer related genetic changes in the tumor. Optional: This clinical trial will conduct extra imaging studies for research purposes including combined endorectal prostate magnetic resonance imaging (MRI), magnetic resonance spectroscopy (MRSI) and diffusion weighted imaging (DWI) to evaluate prostate cancer and response to study treatment.

ELIGIBILITY:
Patients must have newly diagnosed prostate cancer with at least one of the following criteria:

* Clinical Stage > T2
* PSA > 15 ng/ml
* Biopsy Gleason's sum > 8
* All patients must have a minimum PSA value of > 5 ng/ml.
* Patients may not have evidence of distant systemic metastasis.
* Patients may not undergo concurrent hormonal, biologic, or chemotherapy.
* Patients may not have prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil.
* Patients with a history of severe reaction to docetaxel or other drugs formulated with polysorbate 80 will not be eligible.
* Patients may not have an underlying cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-03; Primary Completion 2005-01 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who respond to treatment | 6 months
  To evaluate the response rate associated with capecitabine and docetaxel combination chemotherapy in selected patients with localized or locally advanced prostate cancer. Response is defined as a reduction in the PSA (Prostate Specific Antigen) by at least 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hussain, MD, Principal Investigator — The University of Michigan Comprehensive Cancer Center
Locations (2):
- United States (2):
  - The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan